CLINICAL TRIAL: NCT04327167
Title: Digital Intervention for Ethnic Groups in Transplantation (DIGIT)
Acronym: DiGiT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRAS 250798
Record Dates: First submitted 2019-12-03; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Live Donors, Ethnic Minorities, Transplantation
MeSH Terms: interventions — Videotape Recording; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital intervention (Other)
  Interventions: Behavioral: Video and questionnaire

INTERVENTIONS:
Behavioral: Video and questionnaire — Potential donors would be shown a video and asked to complete a questionnaire to capture change in attitude towards donation.
  Other Names: Digital intervention

SUMMARY:
Study Title Digital intervention for Ethnic Groups in Transplantation (DiGiT)

Internal ref. no. (or short title) DiGiT Study Design Observational cohort study Study Participants 90 Planned Size of Sample (if applicable) 30 Follow up duration (if applicable) 2 years Planned Study Period 2 years Research Question/Aim(s)

1. To produce, test and pilot a video-based intervention about living donor kidney transplantation in Black, Asian & Minority ethnic (BAME) community in United Kingdom. Embedded within this is an ambassador training.
2. Study the long term psychological impact of BAME donors following donation.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Belong to a BAME community only for phase 1-3, in phase 4 all past and future donors regardless of ethnicity would be eligible.
* Be a community member, past donor, past recipient of a transplant, healthcare professional or be on the waiting list for a transplant.

Exclusion Criteria:

* Anyone less than 18 years of age
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the change in score assessing knowledge of LDKT by study questionnaire | 2 years
  Change in attitudes and knowledge of LDKT will be assessed by study questionnaire and the magnitude in change will be quantified by the change in score following digital intervention

SECONDARY OUTCOMES:
Magnitude of change in QOL score pre donation to 1 year post donation | 2 years
  Change in QOL as measured by SF 36 in the 3 months preceding donation and 1 year post donation.

CONTACTS AND LOCATIONS:
Locations (1):
- Shafi Malik, Coventry, West Midlands, United Kingdom

REFERENCES:
- [Derived] Brand S, Daga S, Mistry K, Morsy M, Bagul A, Hamer R, Malik S. Sikh and Muslim perspectives on kidney transplantation: phase 1 of the DiGiT project - a qualitative descriptive study. BMJ Open. 2023 Dec 1;13(12):e059668. doi: 10.1136/bmjopen-2021-059668. PMID 38040423